CLINICAL TRIAL: NCT01837433
Title: Efficiency and Safety Study of Short-term Prednisone to Treat Moderate and Severe Subacute Thyroiditis
Brief Title: Short-term Prednisone to Treat STA Study(SPTSS)
Acronym: STA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Lian Duan, Clinical Doctor, Xinqiao Hospital of Chongqing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XinqiaoH-001
Record Dates: First submitted 2013-04-06; First posted 2013-04-23 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Subacute Thyroiditis
Keywords: Efficacy; safety; short; term; subacute thyroiditis
MeSH Terms: conditions — Thyroiditis, Subacute | interventions — Prednisone; Glucocorticoids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prednisone 1 week (Experimental): Prednisone 1 week 30mg/day and Celecoxib 400mg in first day, and then 200mg bid in the remaining next week, total 2 weeks.
  Interventions: Drug: Prednisone 1 week
- Prednisone 6 weeks (Active Comparator): Oral 30 mg/day of prednisone will be administered as the initial dose for the treatment of SAT in first week,then tapered by 5mg every 1 week,the duration of prednisone will be 6 weeks.
  Interventions: Drug: Prednisone 6 weeks

INTERVENTIONS:
Drug: Prednisone 1 week — Prednisone 1 week 30mg/day and Celecoxib 400mg in first day, and then 200mg bid in the remaining next week, total 2 weeks.
  Other Names: Glucocorticoid
  Arms: Prednisone 1 week
Drug: Prednisone 6 weeks — Guidelines recommend
  Other Names: Glucocorticoid
  Arms: Prednisone 6 weeks

SUMMARY:
Efficiency and Safety Study of Short-term Prednisone to Treat Moderate and Severe Subacute Thyroiditis

The investigators hypothesize that less adverse reactions will be observed, comparing with the guidelines recommend. The recurrence rate, adrenal insufficiency, temporary and permanent hypothyroidism aren't significant difference.

DETAILED DESCRIPTION:
Comparing with the guidelines recommend, short-term (one week)prednisone and nsaids following up next week to treat moderate and severe subacute thyroiditis will be assessed.

The patients in wards will be assessed from temperature,erythrocyte sedimentation rate,C-reactive protein,local pain and goiter.The random treatment will be executed in moderate and severe SAT after informed consent be signed.

Subjects will be monitored once every 2 weeks.If patients complained of pain in their neck or if the erythrocyte sedimentation rate is still high,after discontinuation of prednisone, prednisone treatment will be resumed in moderate and severe subject and non-steroidal anti-inflammatory drugs will be used in mild subject.Anti-ulcer drugs will be administered to all patients.

The endpoint of the study are efficiency and safety of short-term prednisone treating. The investigators will assess adrenal insufficiency (such as anorexia, nausea, vomiting, abdominal pain),steroid withdrawal syndrome, recurrence rate and hypothyroidism. The investigators will observe erythrocyte sedimentation rate,pain,steroid level and thyroid function.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years patients with Moderate and severe subacute thyroiditis

Exclusion Criteria:

* adrenal cortical dysfunction,
* use of corticosteroids in nearly three months,
* mild subacute thyroiditis,
* non-onset STA,
* family history of diabetes,
* gastric ulcer,
* the special medication history,
* heart，liver and renal insufficiency,
* tumors,
* tuberculosis and
* poor compliance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The Efficiency of experimental group comparing with control group during 14 days | 14 days
  We will observe change of erythrocyte sedimentation rate from >20mm/h to normal,C-reactive protein,pain and goiter disappear after 14 days.

SECONDARY OUTCOMES:
recurrence rate | 180 days
  The recurrence will be defined:local tenderness, goiter, inflammatory factors such as erythrocyte sedimentation rate, C-reactive protein increased during 180 days.
hypothyroidism | 180 days
  change in thyroid function:from hyperthyroidism on baseline to hypothyroidism after 180 days.
Adrenal insufficiency after withdraw in experimental group and control group. | 42 days
  The Symptom such as anorexia, nausea, vomiting, abdominal pain, fatigue, weakness, collapse, muscle pain, joint pain, weight loss, orthostatic hypotension, lethargy and depression.
Change of blood glucose in experimental group and control group. | 42 days
  Glucose change when taking medicine:from normal blood glucose on baseline to hyperglycemia at the special time during medication.
Change of blood pressure in experimental and control group during medication. | 42 days
  We will measure blood pressure before and after withdraw prednisone in experimental and control group.
Bone metabolism after withdraw in experimental group and control group. | 42 days
  We will measure Bone metabolism markers before and after withdraw prednisone in experimental and control group.
Change of Lipids in experimental and control group during medication. | 42 days
  We will measure Lipids before and after withdraw prednisone in experimental and control group.

OTHER OUTCOMES:
Other side effects of prednisone | 42 days
  Such as,cushing appearance; female hirsutism, menstrual disorders, impotence in men; gastrointestinal ulcers; psychiatric symptoms: anxiety, agitation, fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Hongting Zheng, Ph.D, Principal Investigator — Department of Endocrinology, The Second Affiliated Hospital, Third Military Medical University, Chongqing, People's Republic of China.
Locations (1):
- The Second Affiliated Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Result] Kubota S, Nishihara E, Kudo T, Ito M, Amino N, Miyauchi A. Initial treatment with 15 mg of prednisolone daily is sufficient for most patients with subacute thyroiditis in Japan. Thyroid. 2013 Mar;23(3):269-72. doi: 10.1089/thy.2012.0459. PMID 23227861
- [Result] Fatourechi V, Aniszewski JP, Fatourechi GZ, Atkinson EJ, Jacobsen SJ. Clinical features and outcome of subacute thyroiditis in an incidence cohort: Olmsted County, Minnesota, study. J Clin Endocrinol Metab. 2003 May;88(5):2100-5. doi: 10.1210/jc.2002-021799. PMID 12727961
- [Result] Nishihara E, Ohye H, Amino N, Takata K, Arishima T, Kudo T, Ito M, Kubota S, Fukata S, Miyauchi A. Clinical characteristics of 852 patients with subacute thyroiditis before treatment. Intern Med. 2008;47(8):725-9. doi: 10.2169/internalmedicine.47.0740. Epub 2008 Apr 16. PMID 18421188
- [Result] Bahn Chair RS, Burch HB, Cooper DS, Garber JR, Greenlee MC, Klein I, Laurberg P, McDougall IR, Montori VM, Rivkees SA, Ross DS, Sosa JA, Stan MN; American Thyroid Association; American Association of Clinical Endocrinologists. Hyperthyroidism and other causes of thyrotoxicosis: management guidelines of the American Thyroid Association and American Association of Clinical Endocrinologists. Thyroid. 2011 Jun;21(6):593-646. doi: 10.1089/thy.2010.0417. Epub 2011 Apr 21. PMID 21510801
- [Result] Nishihara E, Amino N, Ohye H, Ota H, Ito M, Kubota S, Fukata S, Miyauchi A. Extent of hypoechogenic area in the thyroid is related with thyroid dysfunction after subacute thyroiditis. J Endocrinol Invest. 2009 Jan;32(1):33-6. doi: 10.1007/BF03345675. PMID 19337012
- [Result] Iitaka M, Momotani N, Ishii J, Ito K. Incidence of subacute thyroiditis recurrences after a prolonged latency: 24-year survey. J Clin Endocrinol Metab. 1996 Feb;81(2):466-9. doi: 10.1210/jcem.81.2.8636251.
- [Result] Vagenakis AG, Abreau CM, Braverman LE. Prevention of recurrence in acute thyoiditis following corticosteroid withdrawal. J Clin Endocrinol Metab. 1970 Dec;31(6):705-8. doi: 10.1210/jcem-31-6-705. No abstract available. PMID 4098399
- [Result] Volpe R. The management of subacute (DeQuervain's) thyroiditis. Thyroid. 1993 Fall;3(3):253-5. doi: 10.1089/thy.1993.3.253. PMID 8257868
- [Result] Pearce EN, Farwell AP, Braverman LE. Thyroiditis. N Engl J Med. 2003 Jun 26;348(26):2646-55. doi: 10.1056/NEJMra021194. No abstract available. PMID 12826640
- [Result] Desailloud R, Hober D. Viruses and thyroiditis: an update. Virol J. 2009 Jan 12;6:5. doi: 10.1186/1743-422X-6-5. PMID 19138419
- [Result] Mizukoshi T, Noguchi S, Murakami T, Futata T, Yamashita H. Evaluation of recurrence in 36 subacute thyroiditis patients managed with prednisolone. Intern Med. 2001 Apr;40(4):292-5. doi: 10.2169/internalmedicine.40.292. PMID 11334386
- [Result] Benbassat CA, Olchovsky D, Tsvetov G, Shimon I. Subacute thyroiditis: clinical characteristics and treatment outcome in fifty-six consecutive patients diagnosed between 1999 and 2005. J Endocrinol Invest. 2007 Sep;30(8):631-5. doi: 10.1007/BF03347442. PMID 17923793
- [Result] Carella MJ, Srivastava LS, Gossain VV, Rovner DR. Hypothalamic-pituitary-adrenal function one week after a short burst of steroid therapy. J Clin Endocrinol Metab. 1993 May;76(5):1188-91. doi: 10.1210/jcem.76.5.8388401.
- [Result] Alves C, Robazzi TC, Mendonca M. Withdrawal from glucocorticosteroid therapy: clinical practice recommendations. J Pediatr (Rio J). 2008 May-Jun;84(3):192-202. doi: 10.2223/JPED.1773. PMID 18535733
- [Result] Krasner AS. Glucocorticoid-induced adrenal insufficiency. JAMA. 1999 Aug 18;282(7):671-6. doi: 10.1001/jama.282.7.671. No abstract available. PMID 10517721
- [Result] Henzen C, Suter A, Lerch E, Urbinelli R, Schorno XH, Briner VA. Suppression and recovery of adrenal response after short-term, high-dose glucocorticoid treatment. Lancet. 2000 Feb 12;355(9203):542-5. doi: 10.1016/S0140-6736(99)06290-X. PMID 10683005
- [Result] Longui CA. Glucocorticoid therapy: minimizing side effects. J Pediatr (Rio J). 2007 Nov;83(5 Suppl):S163-77. doi: 10.2223/JPED.1713. Epub 2007 Nov 14. PMID 18000630